CLINICAL TRIAL: NCT05770024
Title: Defining, Evaluating, and Sharing Methodologies for Quality Control in Diagnostic Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS SYNLAB SDN (Other)
Responsible Party: Sponsor
Other Study IDs: 10/20
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-03

CONDITIONS: Subjects Undergoing Diagnostic Imaging Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: imaging tests — X-ray radiography (RX); computer tomography (CT); magnetic resonance (MR); positron emission tomography (PET); single photon emission computed tomography (SPECT)

SUMMARY:
The purpose of the study is to validate a radiological quality control (QC) system on the performance of diagnostic imaging. Patient images, previously anonymized by each radiologic diagnostic structures (SDR), will be sent to the QC service, which will blindly submit the images for evaluation external peer review by experts in the field. Through the blinded approach, the information obtained from the QC will allow the SDR to know its own performance analytics, but not those of other SDRs using the service, and to a centralized system to have an anonymized estimate of the quality of performance delivered. Finally, the analyzed data will provide not only a mere count, but will allow to reduce and prevent errors in the appropriateness, execution, reporting and diagnostic content of the examinations

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic examinations related to imaging modalities (RX, CT, MR, PET, SPECT...), agreed with SDRs, of body districts on which diagnostic images are available in DICOM format, medical history data and clinical question, report

Exclusion Criteria:

* Incompleteness of data for the purpose of the review process

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing diagnostic imaging tests
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Definition and implementation of diagnostic image quality control procedures for the purpose of purposes of monitoring the accuracy and appropriateness of the service provided by SDRs | 1-36 months
  * Definition of a survey for evaluation of diagnostic procedures;
  * Definition of a panel of experts;
  * Optimization of radiological quality control workflow;
  * Identification of elements for workflow automation;
  * Definition of feedback strategies for the improvement of procedures diagnostics

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Synlab SDN, Naples, Italy